CLINICAL TRIAL: NCT02773784
Title: Comparison of Core Needle Biopsy (CNB) and Surgical Specimens for Estrogen Receptor (ER), Progesterone Receptor (PgR), Human Epidermal Growth Factor Receptor 2 (HER2) Status and Ki67 Index in Invasive Breast Cancer.
Brief Title: Comparison of CNB and Surgical Specimens for ER, PgR, HER2 Status and Ki67 Index in Invasive Breast Cancer.
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Director of Breast Center of Peking University Cancer Hospital, Peking University
Other Study IDs: BCP16
Record Dates: First submitted 2015-09-16; First posted 2016-05-16 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Invasive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ER, PgR, Her-2 and Ki67 are determined by immunohistochemistry (IHC) in CNB and surgical specimen. FISH analysis will be carried out in all HER2 2+ samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- invasive breast cancer: Patients with invasive breast cancer diagnosed by core needle biopsy (CNB) and not to receive neoadjuvant system therapy are eligible for this study. ER, PR, Her-2 and Ki67 are determined by immunohistochemistry (IHC) in CNB and surgical specimen. FISH analysis will be carried out in all HER2 2+ samples.
  Interventions: Other: immunohistochemistry and/or FISH

INTERVENTIONS:
Other: immunohistochemistry and/or FISH — Patients with invasive breast cancer diagnosed by core needle biopsy (CNB) and not to receive neoadjuvant system therapy are eligible for this study. ER, PR, Her-2 and Ki67 are determined by immunohistochemistry (IHC) in CNB and surgical specimen. FISH analysis will be carried out in all HER2 2+ samples.

SUMMARY:
* This is a prospective, single-center, non-randomized, non-controlled study.
* The estrogen receptor (ER), progesterone receptor (PgR), HER2 status and Ki67 index of CNB specimen are critical biomarkers for making neoadjuvant therapy strategy in invasive breast cancer. The concordance of these biomarkers between CNB and surgical specimen was varied in previous retrospective reports. The aim of this study is to determine the discordance of these biomarkers between CNB and surgical specimen and the influence of making treatment strategy by the discordance.

ELIGIBILITY:
Inclusion Criteria:

* • histologically confirmed primary invasive breast cancer by core needle biopsy

Exclusion Criteria:

* • pathological diagnosed ductal carcinoma in situ or microinvasive breast cancer by core needle biopsy

  * patient plans to receive neo-adjuvant system therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: invasive breast cancer diagnosed by core needle biopsy
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The accuracy of ER, PgR, Her-2 and Ki67 for core needle biopsy (CNB) using the surgical specimens as reference, respectively. | within 4 weeks after obtaining the post-surgery pathological results
  The accuracy of ER, PgR, Her-2 and Ki67 for core needle biopsy (CNB) will be assessed by four parameters respectively, which are sensitivity, specificity, the negative predictive values and the positive predictive values, using the surgical specimens as reference.

SECONDARY OUTCOMES:
Discordance of system therapy strategies between using biomarkers of CNB and surgical specimens. | within 4 weeks after obtaining the post-surgery pathological results

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-Qing Fan, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China